CLINICAL TRIAL: NCT06430099
Title: Rate of Blood Pressure Control Among Hypertensive Patients With Hemodialysis in Sohag University Hospital
Status: Not yet recruiting | Type: Observational
Sponsor: Hager Abdo Mohamed (Other)
Responsible Party: Sponsor-Investigator, Hager Abdo Mohamed, Principal Investigator, Sohag University
Organization: Sohag University (Other)
Other Study IDs: Sohagu.
Record Dates: First submitted 2024-05-21; First posted 2024-05-28 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Hemodialysis; Hypertension
Keywords: hypertension hemodialysis
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this Cross-sectional study is to detect hypertensive patients with hemodialysis in Sohag University Hospital and controlled patients and noncontrolled patients. The main questions it aims to answer are:

1. What is the pattern of blood pressure control among patients receiving hemodialysis?
2. What are factors associated with successful blood pressure control?
3. What is the level of patient knowledge and awareness regarding blood pressure management?
4. What are the challenges and barriers faced by patients in achieving optimal blood pressure control? Participants Blood pressure calculated by taking the average of three consecutive days measurement.

DETAILED DESCRIPTION:
1. Survey Type: Cross-sectional study.
2. Target Population: Patients undergoing hemodialysis.
3. Sample Size: The target sample size are all hypertensive patients in Sohag university hospital dialysis unit
4. Survey Method: person to person interview in dialysis units will be used for data collection.

Blood pressure calculated by taking the average of three consecutive days

* 1st day (Dialysis Day): - Blood pressure will be measured (pre dialysis, inter dialysis, post dialysis).
* 2nd day (Inter Dialytic Day): - Blood pressure will be measured two times (AM, PM).
* 3rd day (Dialysis Day): - Blood pressure will be measured (pre dialysis, inter dialysis, post dialysis).

ELIGIBILITY:
Inclusion Criteria:

- Participants must be

* 18 years or older.
* currently receiving hemodialysis.
* Hypertensive patients.

Exclusion Criteria:

* patients under 18 years old.
* Patients stopped hemodialysis.
* Patients with ESRD not receiving hemodialysis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: hypertensive patients with hemodialysis in Sohag University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-05-24 (Estimated); Primary Completion 2024-12-20 (Estimated); Study Completion 2024-12-20 (Estimated)

PRIMARY OUTCOMES:
Rate of blood pressure control among hypertensive patients with hemodialysis in Sohag University Hospital with hemodialysis in Sohag University Hospital | 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Hassan A Hassanien, professor, Study Chair — Sohag University; Alaa A Ghaleb, professor, Study Chair — Sohag University; Ahmed N Nour Eldin, Lecturer, Study Chair — Sohag University
Locations (1):
- Faculty of Medicine Sohag University, Sohag, Egypt

REFERENCES:
- [Background] Susel J, Batycka-Baran A, Reich A, Szepietowski JC. Uraemic pruritus markedly affects the quality of life and depressive symptoms in haemodialysis patients with end-stage renal disease. Acta Derm Venereol. 2014 May;94(3):276-81. doi: 10.2340/00015555-1749. PMID 24217858
- [Background] Lopes AA, Bragg J, Young E, Goodkin D, Mapes D, Combe C, Piera L, Held P, Gillespie B, Port FK; Dialysis Outcomes and Practice Patterns Study (DOPPS). Depression as a predictor of mortality and hospitalization among hemodialysis patients in the United States and Europe. Kidney Int. 2002 Jul;62(1):199-207. doi: 10.1046/j.1523-1755.2002.00411.x. PMID 12081579
- [Background] Joshi VD. Quality of life in end stage renal disease patients. World J Nephrol. 2014 Nov 6;3(4):308-16. doi: 10.5527/wjn.v3.i4.308. PMID 25374827
- [Background] Garcia-Llana H, Remor E, Selgas R. Adherence to treatment, emotional state and quality of life in patients with end-stage renal disease undergoing dialysis. Psicothema. 2013 Feb;25(1):79-86. doi: 10.7334/psicothema2012.96. PMID 23336548